CLINICAL TRIAL: NCT05940012
Title: Specific and Shared Mechanisms Associated With Physical Therapy Interventions
Brief Title: Specific and Shared Mechanisms Associated With Treatment for Chronic Neck Pain
Acronym: SS-MECH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Saint-Joseph University (Other); Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO00113663
Record Dates: First submitted 2023-05-26; First posted 2023-07-11 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2024-11

CONDITIONS: Chronic Neck Pain
MeSH Terms: interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant
Masking Description: Subjects are told they will be randomized into two forms of treatment for chronic neck pain and that the study team is interested in learning the mechanisms associated with that treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual therapy treatment (Experimental): Manual therapy treatments will consist of global soft tissue stretching of the upper trapezius, occipital muscles, levator scapula, and scalene muscles as the patient lies in supine. Non-thrust manipulation will consist of unilateral or central posterior-anterior accessory movements (PAIVMs) to the cervical and upper thoracic segments (in prone) at the most symptomatic levels. Passive physiological intervertebral movements of rotation will be performed in supine, as a mechanism to reduce pain and increase range of motion. Individuals with chronic neck pain randomized to the manual therapy arm, will be assigned a HEP twice daily that will consist of cervical rotations with belt or equivalent, side flexion with belt or equivalent, self-stretching exercises that are designed to target the upper thoracic musculature, and corner wall stretches.
  Interventions: Other: Manual Therapy
- Resisted exercise treatment (Active Comparator): In-clinic exercises will consist of chin retractions in sitting, supine clock isometric resistance, supine anterior neck flexion exercises that target the deep neck flexors, prone neck extensor exercises (with concurrent chin retraction), and lateral neck raises (bilaterally). The study team will also target the mid and upper thoracic region by performing upright rows, supine chest raises that target the mid-scapular muscles and the paraspinal muscles, prone "I, T, and Y" exercises, and proprioceptive neuromuscular facilitation exercises using a bar or a cane. Individuals randomized to the resistance exercise arm will be assigned a HEP twice daily that will consist of chin retractions in sitting, supine anterior neck flexion exercises, and elastic band rows that replicate the upright rows performed in the clinic.
  Interventions: Other: Manual Therapy

INTERVENTIONS:
Other: Manual Therapy — Hands on treatments including manipulation, mobilization and soft-tissue mobilization with therapeutic intent.
  Other Names: Force based manipulations

SUMMARY:
It is expected that different physical therapy treatments influence outcomes in many different ways. Each treatment is assumed to have a "specific" treatment mechanism, which explains how that specific treatment works. Different treatments also have "shared" mechanisms, which are similar across many different types of interventions (e.g., exercise, cognitive treatments or manual therapy). In this study, the study team will investigate the several types of specific treatment mechanisms of a manual therapy-based approach and an exercise-based approach and the study team will compare these to see if they are different. The patient population will include individuals with chronic neck pain, which is a condition that leads to notable disability and pain. The study team will also evaluate several shared treatment mechanisms to see if these are similar across the two treatments (e.g., manual therapy versus exercise). The study team expects to find that there are some specific treatment mechanisms with each approach (manual therapy versus exercise) but also several "shared" mechanisms that are similar across the two seemingly different approaches. These will likely influence the outcomes and may help explain why clinicians see similar outcomes across both treatment groups for chronic neck pain. This study is important because no one has investigated whether the outcomes that occur with chronic neck pain are mostly influenced by specific or shared treatment mechanisms. Interestingly, in the psychological literature, shared treatment mechanisms demonstrate the strongest influence (more than specific treatment mechanisms).

DETAILED DESCRIPTION:
Treatment mechanisms involve the steps or processes through which an intervention unfolds and produces the change in an outcome variable. In other words, a treatment mechanism is "how a treatment works". Treatment mechanisms can be specific to the intervention provided (i.e., fiber size increase and neuro adaptation occur with resistance exercise) or shared with other treatments (i.e., theoretically, increased therapeutic alliance and reduced fear of movement occur with almost all forms of interventions). In this proposal, the study team plans to investigate specific and shared treatment mechanisms of a manual therapy approach and a resistance exercise approach for treatment of chronic neck pain. The study team is targeting chronic neck pain because it is a common problem that is second only to low back pain for years lived with disability. Routinely, chronic neck pain management includes manual therapy and resistance exercise, as both approaches are included in clinical practice guidelines. The study plans to answer two research questions: 1) what are the specific mechanisms associated with manual therapy and resistance exercise interventions (and are these different), and 2) what are the shared mechanisms associated with these interventions, and do both mechanisms mediate clinical outcomes? The study team hypothesized that manual therapy and resistance exercise approaches will exhibit different specific treatment mechanisms. Further, the team hypothesizes that both approaches will lead to shared treatment mechanisms, which will notably influence outcomes at both 4 weeks and 6-month follow-up. This study is important because it will help identify how different treatment mechanisms influence clinical outcomes. There are several studies in the psychological literature that demonstrate the role of both specific and shared treatment mechanisms but this form of investigation is mostly absent for general musculoskeletal rehabilitation interventions. It will be the first study involving manual therapy in which specific and shared mechanisms are evaluated and explored against clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with chronic neck pain (chronic pain is defined using the International Association of the Study of Pain (IASP) pragmatic criteria of pain lasting for 3 months or more that cannot be attributed to another diagnosis or condition.)
* 18 years of age and older
* experience ongoing neck pain of ≥3 on a 10-point scale for most days of the previous 3-months.

Exclusion Criteria:

* Individuals with cervical pain and suspected radicular symptoms
* a history of neck surgery within 1 year
* current or suspected red flags
* unable to speak or write in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-10-22 (Actual)

PRIMARY OUTCOMES:
Changes in Cervical Range of motion device (CROM) in flexion using a CROM | Baseline, 2 weeks, and 3 weeks
Changes in Cervical Range of motion device in extension using a CROM | Baseline, 2 weeks, and 3 weeks
Changes in Cervical Range of motion device rotation using a CROM | Baseline, 2 weeks, and 3 weeks
Changes in Cervical Range of motion device in side flexion using a CROM | Baseline, 2 weeks, and 3 weeks
Changes in Pain Pressure Threshold with Algometry | Baseline, 2 weeks, and 3 weeks
Changes in time held with the Deep Neck Flexor Endurance Test | Baseline, 2 weeks, and 3 weeks
Changes in in time held with the Cervical Extensor Endurance Test | Baseline, 2 weeks, and 3 weeks
Changes in in time held with the Lateral Neck Flexor Endurance Test for left side | Baseline, 2 weeks, and 3 weeks
Changes in in time held with the Lateral Neck Flexor Endurance Test for right side | Baseline, 2 weeks, and 3 weeks

SECONDARY OUTCOMES:
Change in the Working Alliance Inventory (WAI). | Baseline, 2 weeks and 3 weeks
  The WAI evaluates the collaborative relationship between the helper and the client, but does not encompass all aspects of the therapy relationship (i.e. clinical outcomes, recidivism).The WAI is a 36 item scale with 3 domains (task, goal and bond). Each item is scored 1 to 7, with higher scores reflecting better alliance with the therapist. Total scores range from 36 (low alliance) to 252 (higher alliance). Higher scores are better.
Change in the the OSPRO-YF-10 | Baseline, 2 weeks and 3 weeks
  The OSPRO-YF is a 10 item Optimal Screening for Prediction of Referral and Outcome cohort yellow flag assessment tool. As OSPRO-YF summarizes 11 psychological questionnaires, it is not scored like a conventional screening tool. Quartile scores are used instead of cutoff scores for consistency and assessment of a wide range of outpatient orthopedic patients. Scores that are in the top quartile (top 25%) for negative psychological questionnaires (Negative Mood and Fear Avoidance questionnaires). Scores that are in the bottom quartile (bottom 25%) for positive psychological questionnaires (Positive Affect/Coping questionnaires).
Change in the University of Washington Pain-Related Self Efficacy Scale short form | Baseline, 2 weeks and 3 weeks
  The UW Pain Related Self-Efficacy Scale is intended for measuring disability management self-efficacy in adults with chronic health conditions. The 6 items on the short form are summed using the values provided for each response available in the clinician/researcher version of the form. This will give a summary score that ranges from 6 to 30. Using the Summary Score to T-score Conversion Table, we will use the summary score to look up the IRT-based T-score in the column labeled "Tscore" in the conversion table (page 7 below). This T-score is the final score we will use for all analyses.
Change in Patient Health Engagement Scale | Baseline, 2 weeks and 3 weeks
  The Patient Health Engagement Scale (PHE-s) is a patient self-administrable short psycho-metric questionnaire developed with the aim of diagnosing the level of patient engagement in their healthcare process that is function of his/her degree of emotional elaboration of the health condition. The scale has six items and each item is scored 1 to 7. A low score is poorer engagement whereas a higher score reflects higher engagement. Scores range from six to 42.
Change in the PROMIS 29.2. | Baseline, 4 weeks, and 6 months
  The PROMIS-29 v2.0 profile assesses pain intensity using a single 0-10 numeric rating item and seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance) using four items per domain. Pain intensity is measured 0 to 10, with higher scores reflecting more pain. The other scales are measured as a t score, where 50% reflects the norm and value lower or higher reflect the current scoring by standard deviation to the general population.

CONTACTS AND LOCATIONS:
Overall Officials: Chad E Cook, Principal Investigator — Duke University
Locations (1):
- The Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
The proposal will follow the data sharing guidelines set forth for the NIH HEAL Initiative®. As with the HEAL initiative, we plan to create an infrastructure that addresses the need for researchers, clinicians, and patients to collaborate on sharing their collective data. Our Data Sharing Plan that (1) will make the two projected Publications Open Access and, to the extent possible, and (2) will make the Underlying Primary Data immediately and broadly available to the public. Underlying Primary Data should be made as widely and freely available as possible while safeguarding the privacy of participants and protecting confidential and proprietary data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Protocol when published. SAP within the protocol when published. Informed consent once approval of IRB.